CLINICAL TRIAL: NCT06169657
Title: Comparison of Intensity and Step Count of Gait Training Modalities in the Inpatient Rehabilitation Setting in Sub-acute Central Nervous System Injury
Brief Title: Comparison of Gait Training Methods in Sub-acute Stroke and Spinal Cord Injury
Status: Withdrawn | Type: Observational
Why Stopped: The study team had been practicing running the study interventions, but the core study team members left the organization before any subjects could be enrolled. There is now insufficient personnel time dedication to this study, so it is being closed.
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00219486
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Incomplete Spinal Cord Injury
Keywords: Stroke; Incomplete Spinal Cord Injury; Gait Rehabilitation; Exoskeleton; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Inpatients Post-stroke, low level ambulators: Individuals post acute or subacute stroke that that are inpatients at the Shirley Ryan AbilityLab ages 18-75 with initial gait speed 0.0-0.39 m/s
  Interventions: Device: Body-weight-supported treadmill training (BWSTT); Device: EksoNR exoskeleton gait training; Device: Overground gait training
- Inpatients Post-stroke, high level ambulators: Individuals post acute or subacute stroke that that are inpatients at the Shirley Ryan AbilityLab ages 18-75 with initial gait speed 0.4-0.79 m/s
  Interventions: Device: Body-weight-supported treadmill training (BWSTT); Device: EksoNR exoskeleton gait training; Device: Overground gait training
- Inpatients with iSCI, low level ambulators: Individuals post-SCI or subacute that that are inpatients at the Shirley Ryan AbilityLab ages 18-75 with initial gait speed 0.0-0.39 m/s
  Interventions: Device: Body-weight-supported treadmill training (BWSTT); Device: EksoNR exoskeleton gait training; Device: Overground gait training
- Inpatients with iSCI, high level ambulators: Individuals post-SCI or subacute that that are inpatients at the Shirley Ryan AbilityLab ages 18-75 with initial gait speed 0.4-0.79 m/s
  Interventions: Device: Body-weight-supported treadmill training (BWSTT); Device: EksoNR exoskeleton gait training; Device: Overground gait training

INTERVENTIONS:
Device: Body-weight-supported treadmill training (BWSTT) — Walking on a treadmill in a harness with body weight support as needed
Device: EksoNR exoskeleton gait training — Walking in the EksoNR exoskeleton
Device: Overground gait training — Walking overground in a harness with body weight support as needed

SUMMARY:
The purpose of the project is to compare intensity (minutes in target heart rate zone) and steps per session across three gait training modalities, including body-weight supported treadmill training (BWSTT), overground gait training with body weight-support (BWS), and overground gait training utilizing a lower extremity exoskeleton, between patients presenting with varying functional ambulation capacities in the inpatient setting. Additionally, the researchers will compare physical therapist (PT) burden across these modalities and patient functional presentation levels.

DETAILED DESCRIPTION:
Aim 1 of this study is to measure stepping repetition and intensity via heart rate of three gait-training modalities utilized with patients in the subacute phase of stroke and iSCI during inpatient rehabilitation in order to guide therapists through clinical decision-making of selecting the optimal intervention for patients based on functional presentation. Aim 2 of this study is to measure therapist burden across each gait training modalities, as this is an additional factor that contributes to the number of steps taken and intensity experienced by the patient.

The gait training modalities assessed will include BWSTT, overground gait training with a lower extremity exoskeleton, and overground gait training with BWS. The participants' functional level will be classified by gait speed obtained via the 10 meter walk test (10MWT), a standardized assessment commonly used in rehabilitation. These functional classification categories include household ambulator (low level) and limited community ambulator (high level), determined by Fritz et al. 2009.

The researchers hypothesize that low functioning/household ambulators will achieve more minutes in high-intensity training zones utilizing the exoskeleton due to the enhanced participation and increased weight-bearing the device supports compared to the other modalities. In addition, a greater number steps will be achieved in this mode due to the exoskeleton's ability to decrease overall therapist burden compared to BWSTT and overground with BWS. In contrast, the researchers anticipate that steps per session and overall intensity will be decreased in high functioning/limited community ambulators due the unnecessary support the exoskeleton provides at this functional level. The researchers believe that high functioning/ limited community ambulators will achieve the highest number of steps and intensity during BWSTT due to the ability to increase challenges via treadmill parameters such as speed and incline while utilizing a harness for safety and bodyweight support only as necessary. In contrast, the researchers believe the amount of BWS and assistance a PT must provide relative to the patient's contribution to practice successful stepping during BWSTT will result in a lower intensity and number of steps achieved in low functioning/household ambulators.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, inclusive
* Medical clearance from primary medical team (signed Medical Clearance form)
* Adequate cognitive function as determined by the NIH scale: score ≤1 on question 1b and score =0 on question 1c
* Gait speed between 0-0.79 m/s
* Informed consent provided by participant or POA
* English speaking

Additional Inclusion Criteria for patients post-stroke:

* First stroke, ischemic or hemorrhagic, within the past six months
* Unilateral, supratentorial stroke

Additional Inclusion Criteria for patients iSCI:

* ASIA C or D
* Traumatic iSCI, within past six months

Exclusion Criteria

* Severe aphasia limiting ability to express needs or discomfort verbally or nonverbally
* History of or concurrent neurologic condition (i.e., stroke, SCI, PD, TBI, MS, etc.)
* History of peripheral nerve injury
* Severe knee, hip, or ankle osteoarthritis
* Severe osteoporosis as indicated by physician medical clearance
* Open wounds on skin surfaces in contact with exoskeleton or harness
* Unstable spine or unhealed fractures
* Weight bearing precautions
* Unresolved deep vein thrombosis (DVT)
* Pregnancy
* Prisoners

Additional Exclusion criteria for EksoNR13:

* Weight >220 lbs (100 kg)
* Height below 60 inches or above 76 inches
* Standing hip width of approximately 18 inches or more
* Joint contractures or range of motion deficits that limit normal range of motion during ambulation:

  * Knee flexion contracture greater than 12°
  * Hip flexion contracture greater than 17°
  * Inability to achieve 0° neutral ankle dorsiflexion with knee flexion up to 12°
  * Bilateral hip flexion less than 110°
* Significant spasticity in the lower limbs (Modified Ashworth Scale ≥3)
* Leg length discrepancy:

  * Greater than 0.5 in. (1.27 cm) for upper legs
  * Greater than 0.75 in. (1.91 cm) for lower legs
* Active heterotopic ossification
* Significant spasticity in the lower limbs (Modified Ashworth Scale ≥3)
* High anxiety or claustrophobia
* Clostridium difficile or other gastrointestinal isolation precautions
* Colostomy
* Uncontrolled autonomic dysreflexia
* Lower limb prosthesis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals poststroke or post-iSCI that are inpatients at Shirley Ryan AbilityLab
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-11-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Observation of Step count | Each session through completion of study, up to 10 days
  The number of steps taken during each session will be measured using activity monitors/pedometers. These devices are small accelerometers that can be worn on a belt and/or on the ankle to record steps and Kcals during an activity. The therapist leading the intervention session will apply the ActiGraph at the beginning of each intervention session and remove it upon completion. A higher step count is a better outcome.
Observation of Time spent in age-predicted maximum high-intensity target heart rate zone | Each session through completion of study, up to 10 days
  The target range of 70-85% of age-predicted maximum heart rate will be calculated for each participant utilizing HR max = 208 - [0.7 × age] as developed by Tanka et al in 2001. The target range of 70-85% of age-predicted maximum heart rate will be calculated for each participant. The researchers will record the amount of time participants spend in their pre-calculated target zone during each gait training. The minimum amount of time would be 0 minutes and the maximum amount of time would be 60 minutes as this would be the total time of the session. More time spent in the maximum intensity zone target zone is a better outcome.
Observation of Time spent in age-predicted moderate-intensity target heart rate zone | Each session through completion of study, up to 10 days
  The target range of 50-70% of age-predicted maximum heart rate will be calculated for each participant utilizing HR max = 208 - [0.7 × age] as developed by Tanka et al in 2001. The target range of 50-70% of age-predicted maximum heart rate will be calculated for each participant. The researchers will record the amount of time participants spend in their pre-calculated target zone during each gait training. The minimum amount of time would be 0 minutes and the maximum amount of time would be 60 minutes as this would be the total time of the session. Less time spent in the moderate intensity pre-calculated target zone is a better outcome as the more minutes in the high intensity zone is the best outcome.
Observation of Time spent in age-predicted low-intensity target heart rate zone | Each session through completion of study, up to 10 days
  The target range of 50% of age-predicted maximum heart rate will be calculated for each participant utilizing HR max = 208 - [0.7 × age] as developed by Tanka et al in 2001. Low intensity equals 50% or less of age-predicted maximum heart rate and will be calculated for each participant. The researchers will record the amount of time participants spend in their pre-calculated target zone during each gait training. The minimum amount of time would be 0 minutes and the maximum amount of time would be 60 minutes as this would be the total time of the session. Less time spent in the low intensity zone is better as the goal is to achieve more minutes in high-intensity zone.

SECONDARY OUTCOMES:
Observation of Minutes spent in equipment setup per session | Each session through completion of study, up to 10 days
  Total time in minutes spent applying and removing equipment. The minimum amount of time would be 0 minutes and the maximum amount of time would be 60 minutes as this would be the total time of the session. Less time would be considered better as that indicates more time spent walking.
Observation of Minutes spent in rest breaks per session | Each session through completion of study, up to 10 days
  Total time in minutes the participant spends resting (not walking or applying/ removing equipment) between walking bouts. The minimum amount of time would be 0 minutes and the maximum amount of time would be 60 minutes as this would be the total time of the session. Less time would be considered better as that indicates more time spent walking.
Observation of Minutes spent stepping | Each session through completion of study, up to 10 days
  Total time in minutes the participant spends walking (not including rest breaks or applying/ removing equipment) during a session. The minimum amount of time would be 0 minutes and the maximum amount of time would be 60 minutes as this would be the total time of the session. Less time would be considered better as that indicates more time spent walking.
Observation of Patient Borg Rating of perceived exertion (RPE) | Each session through completion of study, up to 10 days
  The Borg Rating of Perceived Exertion is a tool to measure the subjective report of effort, exertion, and fatigue during physical work. It consists of a 15-point scale from 6-20, in which 6=no exertion and 20=absolute maximum exertion. It is presented to the participant in written format with descriptors to standardize the report of perceived exertion across tasks. An optimal score is between 14-20 as this indicates higher perceived walking intensity for the participant.
Observation of Patient Intrinsic Motivation Inventory (IMI) | Each session through completion of study, up to 10 days
  The Intrinsic Motivation Inventory (IMI) is a multidimensional measurement that measures participants' subjective experience related to a target activity in laboratory experiments. The instrument consists of seven subscale scores related to interest/enjoyment, perceived competence, effort/importance, felt pressure/tension, perceived choice, value/usefulness and relatedness while performing a given activity. 29 items, adapted from the standardized instrument, are addressed on a 7 point scale, 1-7, in which one indicates not at all and seven indicates very true. A higher score is better.
Observation of therapist maximum heart rate | Each session through completion of study, up to 10 days
  Therapist heart rate will be measured throughout each session as an indicator of burden. There is no standard minimum or maximum value, however a higher heart rate indicates increased therapist burden.
Observation of therapist maximum Borg Rating of perceived exertion (RPE) | Each session through completion of study, up to 10 days
  The Borg Rating of Perceived Exertion is a tool to measure the subjective report of effort, exertion, and fatigue during physical work. It consists of a 15-point scale from 6-20, in which 6=no exertion and 20=absolute maximum exertion. It is presented to the participant in written format with descriptors to standardize the report of perceived exertion across tasks. A lower score is better, indicating less burden on the therapist.
Observation of therapist Numerical Pain Rating Scale (NPRS) | Each session through completion of study, up to 10 days
  The NPRS is used to measure the subjective report of pain intensity. It consists of an 11-point scale, 0-10, in which zero indicates no pain and ten indicates the most intense pain imaginable. A lower score is better, indicating less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Pons, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No